CLINICAL TRIAL: NCT01414985
Title: Direct CNS Administration of a Replication Deficient Adeno-associated Virus Gene Transfer Vector Serotype rh.10 Expressing the Human CLN2 cDNA to Children With LINCL With Uncommon Genotypes and/or Moderate to Severe Impairment
Brief Title: AAVRh.10 Administered to Children With Late Infantile Neuronal Ceroid Lipofuscinosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1005011054; IND 13951 (Other: RAC #1008-1064)
Record Dates: First submitted 2010-12-13; First posted 2011-08-11 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Late Infantile Neuronal Ceroid Lipofuscinosis; Batten Disease
Keywords: Batten Disease
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A consists of 2 subjects who received 9x10^11 molecules of AAVrh.10CUCLN2, the gene transfer vector carrying the CLN2 gene. This is equal to 900,000,000,000 molecules of the study drug. The drug will be administered only once in the study.
  Interventions: Biological: AAVrh.10CUCLN2
- Group B (Experimental): Group B will consist of 6 subjects who will receive 2.85x10^11 molecules of AAVrh.10CUCLN2, the gene transfer vector carrying the CLN2 gene. This is equal to 285,000,000,000 molecules of the drug. The drug will be administered only once in the study.
  Interventions: Biological: AAVrh.10CUCLN2

INTERVENTIONS:
Biological: AAVrh.10CUCLN2 — There will be 2 dose cohorts in this study. Group A consists of 2 subjects who have received 9.0x10^11 genome copies (900,000,000,000 molecules) of the study drug, AAVrh.10CUCLN2. Group B will consist of 6 subjects who will receive a lower dose of 2.85x10^11 genome copies (285,000,000,000 molecules) of the study drug, AAVrh.10CUCLN2.
  Other Names: AAVrh.10

SUMMARY:
The investigators propose to assess the safety and efficacy of a new administration method to deliver a biologic to children with a form of Batten disease using an experimental gene transfer procedure. This gene transfer procedure consists of delivering a good copy of the mutated gene to the nerve cells via a virus. These children are born with genetic changes called mutations that result in the inability of the brain to properly recycle proteins. The recycling failure leads to death of the nerve cells in the brain and progressive loss of brain function. Children with Batten disease are normal at birth but by age 2 to 4 have motor and vision problems which progress rapidly to death at age approximately 10 years old. There are no therapies available to treat the disease.

The investigators previous clinical trial used a virus called adeno-associated virus 2 (AAV2) as the gene delivery system. That study showed that viral delivery of the gene was safe and showed small, but significant benefits to the recipient. The investigators currently have an IRB approved protocol which uses a slightly different virus called AAVrh.10 as the gene delivery system. This 3rd protocol proposes to use the same virus AAVrh.10 as the gene delivery system and has expanded the eligibility criteria.

DETAILED DESCRIPTION:
This study is designed to run parallel to our currently IRB approved protocol #0810010013 entitled "Direct CNS Administration of a Replication Deficient Adeno-associated Virus Gene Transfer Vector Serotype rh.10 Expressing the Human CLN2 cDNA to Children with Late Infantile Neuronal Ceroid Lipofuscinosis," which will assess the safety and efficacy of the virus AAVrh.10 to deliver the CLN2 gene to children in the early stages of the disease. This current study proposes to assess the safety and efficacy of the administration of the same biologic to children who do not fit the criteria for IRB protocol #0810010013.

The differences between protocol #0810010013 and the proposed "parallel" protocol is that inclusion criteria have been modified to include children with any genotype (not only the 5 most common genotypes as in the currently approved protocol) and/or those who score below a 6 but at least a 1 on the Weill Cornell LINCL scale. The reason for expanding the eligibility criteria is to obtain a range of safety data for all children with LINCL, not only those with limited genotype and/or severity. Only 8 subjects will be administered the gene transfer vector in this "parallel" protocol. Subjects will be accrued through IRB approved protocol #0901010186 entitled, "Genotype-Phenotype Correlations of Late Infantile Neuronal Ceroid Lipofuscinosis (2)." Those who do not fit all criteria for the already approved gene transfer protocol (#0810010013) may have the opportunity to be enrolled in this proposed "parallel protocol" (Figure 1). The subjects in the new protocol will be compared to the 16 treated and 16 untreated children enrolled in IRB protocol #0810010013 and #0901010186, respectively.

ELIGIBILITY:
Inclusion criteria.

1. Definitive diagnosis of LINCL, based on clinical phenotype and genotype. The study does not limit to one specific genotype (genetic constitution).
2. The subject must be between the age of 3 and 18 years.
3. Subjects will have an average total score of less than 4 but at least 1, and/or an uncommon genotype defined as any genotype that does not include at least one of the 5 most common mutant CLN2 genotypes: C3670T (nonsense Arg208 to stop), G3556C (intron 7 splice), G5271C (Gln422His), T4396G (aberrant splicing, intron8), and G4655A. The total LINCL score should not be outside the 95th percentile confidence limits for age based on our historic data.
4. The subject will not previously have participated in a gene transfer or stem cell study.
5. Parents of study participants must agree to comply in good faith with the conditions of the study, including attending all of the required baseline and follow-up assessments, and both parents or legal guardians must give consent for their child's participation.
6. Sexually active subjects will have to use contraception during the treatment and for 2 months after completion of the treatment.

Exclusion criteria.

1. Presence of other significant medical or neurological conditions may disqualify the subject from participation in this study, particularly those which would create an unacceptable operative risk or risk to receiving the AAVrh.10CUhCLN2 vector, e.g., malignancy, congenital heart disease, liver or renal failure.
2. Subjects without adequate control of seizures.
3. Subjects with heart disease that would be a risk for anesthesia or a history of major risk factors for hemorrhage.
4. Subjects who cannot participate in MRI studies.
5. Concurrent participation in any other FDA approved Investigational New Drug.
6. Subjects with history of prolonged bleeding or abnormal platelet function or taking aspirin.
7. Renal disease or altered renal function as defined by serum creatinine > 1.5 mg/dl at admission.
8. Abnormal serum sodium, potassium calcium, magnesium, phosphate at grade III or IV by Division of AIDS Toxicity Scale
9. Hepatic disease or altered liver function as defined by SGPT > 150 U/L, and or T.Bilirubin> 1.3 mg/dL
10. Immunosuppression as defined by WBC < 3,000 at admission
11. Uncorrected coagulopathy during the baseline period defined as INR > 1.4; PTT > 35 sec; PLT < 150,000/mm3
12. Anemia (hemoglobin < 11.0 mg/dl at > 2 years of age, with normal serum iron studies)

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2010-04-15 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
Change in CNS function, as measured by the Weill Cornell LINCL Scale | Screening, Pre-transfer, Months 1, 6, 12 and 18
  The Weill Cornell LINCL scale, a 12 point scale which combines assessment of feeding, gait, motor and language to give an overall assessment of various CNS functions (Appendix II for the paper describing the scale and Appendix VI for the scale)27. The lowest possible score is 0 (less progressed in disease) and the highest possible score is 12 (more progressed in disease). This rating scale evaluation will be performed by 2 independent pediatricians, on the basis of a videotaped evaluation. If the 2 independent scores differ by 1 or less they will be averaged and if they differ by greater than 1 point, a consensus will be obtained by a 3rd pediatrician. This outcome measure will look at changes over time.
Safety, as measured by MRI | Screening, Pre-transfer, Months 6, 12 and 18
  3 imaging parameters (% gray matter volume, % ventricular volume and cortical apparent diffusion coefficient) correlate with age and the Weill Cornell LINCL scale. These 3 imaging parameters will be used to assess disease progression (control protocol) and safety of the gene transfer vector (vector protocol) over time. In addition to these imaging parameters we will also perform magnetic resonance spectroscopy (MRS) but the data obtained from this will be for information only for method development. This outcome measure will look at changes over time.

SECONDARY OUTCOMES:
Change in Quality of Life, as measured by the Child Health Questionnaire (CHQ) or Infant Toddler Quality of Life (ITQoL) (depending on age) | Screening, Pre-transfer (optional) and Month 18
  The CHQ or ITQoL, a quality of life questionnaire which will be completed by at least one parent/legal guardian at the time of the LINCL patients' visits to Weill Cornell. The survey will be administered independently to each parent to minimize observer bias if both parents are present. This outcome measure looks at a change over time.The lowest possible score is 0 (corresponds to lower health-related quality of life) and the highest possible score is 100 (corresponds to better health-related quality of life).
Change in psychological development, as measured by the Mullen Scale | Screening, Pre-transfer (optional) and Month 18
  The Mullen scale, a pediatric developmental psychological rating scale, will be administered by a developmental psychologist, and be videotaped. This outcome measure will look at changes over time. The lowest possible score is 0 (corresponds to less psychological development) and the highest possible score is 197 (corresponds to better psychological development).

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De BP, Cram S, Lee H, Rosenberg JB, Sondhi D, Crystal RG, Kaminsky SM. Assessment of Residual Full-Length SV40 Large T Antigen in Clinical-Grade Adeno-Associated Virus Vectors Produced in 293T Cells. Hum Gene Ther. 2023 Aug;34(15-16):697-704. doi: 10.1089/hum.2023.032. PMID 37171121